CLINICAL TRIAL: NCT05646849
Title: Using a Connected Application to Maintain Physical Activity After Cardiac Rehabilitation
Acronym: APA&CO2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-A01974-39
Record Dates: First submitted 2022-11-21; First posted 2022-12-12 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Cardiac Rehabilitation; Acute Coronary Syndrome; Heart Failure
Keywords: Cardiac Rehabilitation; Acute Coronary Syndrome; Heart Failure
MeSH Terms: conditions — Acute Coronary Syndrome; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classic care (No Intervention): Home exercise book, personalized advices and development of an individualized project post-cardiac rehabilitation.
- Connected application (Experimental): Recording and sharing sessions. Exchanges and interactions with other patients. Participation in three collective challenges.
  Interventions: Other: Connected application

INTERVENTIONS:
Other: Connected application — Recording and sharing sessions. Exchanges and interactions with other patients. Participation in three collective challenges.
  Arms: Connected application

SUMMARY:
Maintaining physical activity after cardiac rehabilitation has a major role in disease progression and patient prognosis. 6 months after the cardiac rehabilitation, we find during a nursing interview that many patients do not maintain regular physical activity.

1 year after cardiac rehabilitation, between 30% and 60% of patients do not maintain the recommendations in terms of physical activity.

It is recommended to perform studies evaluating the effectiveness of new technologies in the fight against non-compliance recommendations for physical activity.

That is why, study the interest of using an application connected post-cardiac rehabilitation seems necessary to fight against dropouts in terms of physical activity.

DETAILED DESCRIPTION:
The objective is to study compliance with the recommendations, assessed by accelerometer at 6 months post-cardiac rehabilitation within two groups : classic care versus using a connected application.

ELIGIBILITY:
Inclusion Criteria:

* Patient participating in cardiac rehabilitation
* Patient with a smartphone compatible with the application
* Patient with internet connection
* Patient having signed the written consent to participate

Exclusion Criteria:

* Patient reluctant or unable to comply with the protocol
* Pregnant, parturient and nursing mothers
* Persons deprived of their liberty or under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2025-01-11 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
To demonstrate an increase in the percentage of patients respecting at 6 months post-cardiac rehabilitation the recommendations in terms of physical activity | at 6 months
  accelerometer

SECONDARY OUTCOMES:
to study within each group the evolution of the level of physical activity between the end of the cardiac rehabilitation. | at 6 months
  questionnaires IPAQ
to study within each group the evolution of the motivation to physical activity between the end of the cardiac rehabilitation. | at 6 months
  questionnaire EMAPS
to study the difference in the level of physical activity at 6 months post-cardiac rehabilitation between the two groups | at 6 months
  questionnaires IPAQ
to study the difference in the motivation to physical activity at 6 months post-cardiac rehabilitation between the two groups | at 6 months
  questionnaire EMAPS
to describe the maintenance of the physical activity of the two groups according to the seasonality following the end of the cardiac rehabilitation (winter, spring, summer, autumn). | at 6 months
  accelerometer
to describe the use of the application in the intervention group | at 6 months
  number of recorded sessions
to describe patient satisfaction in the intervention group | at 6 months
  scale 0-10 (min 0 - max 10)
to describe the frequency of use of patients in the intervention group to be recorded their sessions | at 6 months
  scale 0-4 (min 0 - max 4)
to describe the interactions with other users in the intervention group | at 6 months
  scale 0-4 (min 0 -max 4)
to describe participation in challenges in the intervention group | at 6 months
  scale 0-3 (min 0 - max 3)
to describe the continued use of the application in the intervention group | at 12 months
  number of recorded sessions
to describe the continued use of the application in the intervention group | at 18 months
  number of recorded sessions

CONTACTS AND LOCATIONS:
Overall Officials: Paul Da Ros Vettoretto, Principal Investigator — Centre Hospitalier de Cholet
Locations (1):
- Ch Cholet, Cholet, France

IPD SHARING:
Plan to Share IPD: No